CLINICAL TRIAL: NCT00230204
Title: Antibodies Screening in Multiple Sclerosis as a Part of an International Survey in Autoimmune Diseases.
Brief Title: Infections and Autoimmunity: Autobodies Screening in Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-05-3868-AA-CTIL
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2006-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Antibodies; Serum; Infectious agents; Immunoglobulin G; Immunoglobulin M
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Procedure: Serum antibodies to infectious agents using the BioPlex 2200 and complementary EIA kits

SUMMARY:
The purpose of this investigation is to assess the prevalence of infectious disease seropositivity (toxoplasmosis, rubella, cytomegalovirus [CMV]), herpes simplex virus type 1 (HSV-1) and herpes simplex virus type 2 (HSV-2), syphilis, Epstein-Barr virus and H. pylori in a group of patients presenting with specific autoimmune diseases (rheumatoid arthritis [RA], undifferentiated connective tissue disorder [UCTD], Sjogren, antiphospholipid syndrome - APS, vasculitides, systemic lupus erythematosus [SLE], polymyositis, Hashimoto, multiple sclerosis, primary biliary cirrhosis [PBC], etc.), using the BioPlex 2200 and complementary EIA kits as compared to matched controls (by age, sex and ethnicity).

DETAILED DESCRIPTION:
The purpose of this investigation is to assess the prevalence of infectious disease seropositivity (toxoplasmosis, rubella, cytomegalovirus [CMV]), herpes simplex virus type 1 (HSV-1) and herpes simplex virus type 2 (HSV-2), syphilis, Epstein-Barr virus and H. pylori in a group of patients presenting with specific autoimmune diseases (RA, UCTD, Sjogren, antiphospholipid syndrome - APS, vasculitides, SLE, polymyositis, Hashimoto, multiple sclerosis, PBC, etc.), using the BioPlex 2200 and complementary EIA kits as compared to matched controls (by age, sex and ethnicity).

We will assess in our Center 100 patients with multiple sclerosis for the antibody profile of different infectious agents. Comparative assessments will be performed with normal matched subjects.

ELIGIBILITY:
Inclusion Criteria:

* Definite multiple sclerosis

Exclusion Criteria:

* Intravenous immune globulin (IVIg) treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2005-09; Study Completion 2006-04

PRIMARY OUTCOMES:
Determine antibodies to infectious agents immunoglobulin G (IgG), IgM in patients with multiple sclerosis

SECONDARY OUTCOMES:
Assess correlation between antibody levels to various infectious agents with clinical disease variables

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, MD, PhD, Principal Investigator — Multiple Sclerosis Center, Sheba Medical Center, Tel-Hashomer, Israel; Yehuda Shoenfeld, Principal Investigator — Center for Autoimmune Diseases, Sheba Medical Center, Tel-Hashomer, Israel
Locations (1):
- Multiple Sclerosis Center, Sheba Medical Center, Ramat Gan, Israel